CLINICAL TRIAL: NCT01092663
Title: The Effects of Co-administration of Colesevelam and Sitagliptin on Glucose Metabolism in Patients With Type 2 Diabetes
Brief Title: The Effects of Co-admin of Colesevelam and Sitagliptin on Glucose Metabolism in Subjects With Type 2 Diabetes Mellitus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KineMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KM-29
Record Dates: First submitted 2010-03-23; First posted 2010-03-25 (Estimated); Results first posted 2013-01-17 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Colesevelam; type 2 diabetes; sitagliptin; glucose metabolism
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Colesevelam Hydrochloride; Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Colesevelam HCl: 3 tablets, 2x/day (Active Comparator): Subjects will be given 3.75 g/day. Subjects will be given 3 tablets (625mg each) with breakfast and 3 tablets (625mg) with dinner for 12 weeks.
  Interventions: Drug: Colesevelam HCl
- Colesevelam plus Sitagliptin (Active Comparator): Colesevelam: Subjects will be given 3.75 g/day. Subjects will be given 3 tablets (625mg each) with breakfast and 3 tablets (625mg) with dinner for 12 weeks.
  Sitagliptin: Subjects will be given 100mg/day. Subjects will be given 1 tablet (100mg) with breakfast for 12 weeks.
  Interventions: Drug: Colesevelam HCl; Drug: Sitagliptin

INTERVENTIONS:
Drug: Colesevelam HCl — Subjects will be given 3.75 g/day. Subjects will be given 3 tablets (625mg each) with breakfast and 3 tablets (625mg) with dinner for 12 weeks.
  Other Names: Welchol
Drug: Sitagliptin — Subjects will be given 100mg/day. Subjects will be given 1 tablet (100mg) with breakfast for 12 weeks.
  Other Names: Januvia
  Arms: Colesevelam plus Sitagliptin

SUMMARY:
This study will assess the effects of colesevelam, alone or in combination with sitagliptin, on glucose metabolism in subjects with T2DM inadequately controlled by diet and exercise

DETAILED DESCRIPTION:
The hypothesis is that co-administrationof colesevelam plus sitagliptin results in a greater reduction in HbA1c compared to colesevelam HCl treatment by

1. improving the effects of colesevelam on fasting glucose metabolism
2. improving the effects of colsevelam on postprandial glucose metabolism

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Females of childbearing potential are on approved birth control method
* Negative pregnancy testing for females of childbearing potential
* Previously diagnosed or newly diagnosed with T2DM drug naïve subjects
* HbA1c: 6.7-10%
* Age 18 - 80 years
* BMI ≥ 18.5 kg/m2 and ≤ 40 kg/m2
* Fasting serum glucose < 300 mg/dL
* Normal liver function, normal thyroid function, no history of liver, biliary or intestinal disease
* Normal TSH
* On stable diet and exercise routine for at least 4 weeks prior to screening
* Has had a stable weight (+/-5%) for ≥3 months before screening

Exclusion Criteria:

* A history of type 1 diabetes mellitus or history of diabetic ketoacidosis
* History of chronic (required daily for > 2 months) use of insulin therapy
* Treatment with blood pressure lowering therapy that has not been stable for three months before screening
* Treatment with lipid lowering medication other than statins
* Treatment with statins that has not been stable for three months before screening
* Treatment with a DPP-4 inhibitor or and GLP1 agonists at any time
* Treatment with a thiazolidinedione (TZD) within the last 6 months of screening
* History of an allergic or toxic reaction to sitagliptin or colesevelam
* History of dysphagia, swallowing disorders, bowel obstruction, intestinal motility disorder, and gastrointestinal disorders
* History of major gastrointestinal surgery
* History of kidney problems
* Fasting plasma triglycerides > 300 mg/dL
* Serum LDL-C <60 mg/dL
* Positive toxicology test
* Known hypersensitivity to colesevelam HCl or sitagliptin.
* Any contraindications to a study medication (colesevelam HCl or sitagliptin).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2010-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carine Beysen, DPhil, Principal Investigator — KineMed, Inc.
Locations (3):
- United States (3):
  - University of California, San Francisco, San Francisco, California
  - Clinical Pharmacology of Miami, Miami, Florida
  - Healthcare Discoveries, LLC d/b/a ICON Development Solutions, San Antonio, Texas

REFERENCES:
- [Background] Zieve FJ, Kalin MF, Schwartz SL, Jones MR, Bailey WL. Results of the glucose-lowering effect of WelChol study (GLOWS): a randomized, double-blind, placebo-controlled pilot study evaluating the effect of colesevelam hydrochloride on glycemic control in subjects with type 2 diabetes. Clin Ther. 2007 Jan;29(1):74-83. doi: 10.1016/j.clinthera.2007.01.003. PMID 17379048
- [Background] Bays HE, Goldberg RB, Truitt KE, Jones MR. Colesevelam hydrochloride therapy in patients with type 2 diabetes mellitus treated with metformin: glucose and lipid effects. Arch Intern Med. 2008 Oct 13;168(18):1975-83. doi: 10.1001/archinte.168.18.1975. PMID 18852398
- [Background] Fonseca VA, Rosenstock J, Wang AC, Truitt KE, Jones MR. Colesevelam HCl improves glycemic control and reduces LDL cholesterol in patients with inadequately controlled type 2 diabetes on sulfonylurea-based therapy. Diabetes Care. 2008 Aug;31(8):1479-84. doi: 10.2337/dc08-0283. Epub 2008 May 5. PMID 18458145
- [Background] Goldberg RB, Fonseca VA, Truitt KE, Jones MR. Efficacy and safety of colesevelam in patients with type 2 diabetes mellitus and inadequate glycemic control receiving insulin-based therapy. Arch Intern Med. 2008 Jul 28;168(14):1531-40. doi: 10.1001/archinte.168.14.1531. PMID 18663165
- [Background] Aschner P, Kipnes MS, Lunceford JK, Sanchez M, Mickel C, Williams-Herman DE; Sitagliptin Study 021 Group. Effect of the dipeptidyl peptidase-4 inhibitor sitagliptin as monotherapy on glycemic control in patients with type 2 diabetes. Diabetes Care. 2006 Dec;29(12):2632-7. doi: 10.2337/dc06-0703. PMID 17130196
- [Background] Nauck MA, Meininger G, Sheng D, Terranella L, Stein PP; Sitagliptin Study 024 Group. Efficacy and safety of the dipeptidyl peptidase-4 inhibitor, sitagliptin, compared with the sulfonylurea, glipizide, in patients with type 2 diabetes inadequately controlled on metformin alone: a randomized, double-blind, non-inferiority trial. Diabetes Obes Metab. 2007 Mar;9(2):194-205. doi: 10.1111/j.1463-1326.2006.00704.x. PMID 17300595
- [Background] Goldstein BJ, Feinglos MN, Lunceford JK, Johnson J, Williams-Herman DE; Sitagliptin 036 Study Group. Effect of initial combination therapy with sitagliptin, a dipeptidyl peptidase-4 inhibitor, and metformin on glycemic control in patients with type 2 diabetes. Diabetes Care. 2007 Aug;30(8):1979-87. doi: 10.2337/dc07-0627. Epub 2007 May 7. PMID 17485570
- See also: Ethics and Compliance — http://www.ich.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study period from February 2010 to December 2010. This was a multi-center, randomized, open-label, prospective, parallel-group study consisting of 12 weeks of active treatment.
Pre-assignment Details: Subjects treated with acarbose, sulfonylurea or metformin and an A1C ≥6.5% and ≤9% were eligible to enter the study after a 4 (acarbose and sulfonylurea) or 8 (metformin) week wash-out period when meeting all other criteria.
Groups:
- Colesevelam: Subjects were given 3.75 g colesevelem per day: 3 tablets (625mg each) with breakfast and 3 tablets with dinner for 12 weeks.
- Colesevelam Plus Sitagliptin: Colesevelam: Subjects were given 3.75 g colesevelem per day: 3 tablets (625mg each) with breakfast and 3 tablets with dinner for 12 weeks.
  Sitagliptin: In addition subjects were given 100mg sitagliptin/day. Subjects were given 1 tablet (100mg) with breakfast for 12 weeks.
Period: Overall Study
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Started | 31 | 30
Completed | 24 | 26
Not Completed | 7 | 4
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Glucose >300mg/dL | 1 | 0
Not completed — High fasting triglyceride | 2 | 0
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Colesevelam: Subjects were given 3.75 g colesevelam per day: 3 tablets (625mg each) with breakfast and 3 tablets (625mg each) with dinner for 12 weeks.
- Total: Total of all reporting groups
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 7 | 9 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (9) | 55 (13) | 55.5 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 26
  Male | 19 | 16 | 35
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 29 | 59
  Not Hispanic or Latino | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 26 | 27 | 53
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 31 | 30 | 61
Weight [Mean (Standard Deviation); unit: kilograms] | 84.6 (15.3) | 85.1 (17.0) | 84.85 (16.15)
BMI [Mean (Standard Deviation); unit: kilograms/square meter (kg/m2)] | 30.7 (3.7) | 30.9 (4.7) | 30.8 (4.2)
Fat Free Mass [Mean (Standard Deviation); unit: kilograms] | 51.4 (10.3) | 54.4 (11.4) | 52.9 (10.85)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage] | 8.0 (0.9) | 8.0 (1.1) | 8.0 (1.0)
Fasting Glucose [Mean (Standard Deviation); unit: millimole/liter (mmol/L)] — glucose measured in the plasma
  millimole/liter (mmol/L) | 8.9 (2.5) | 8.7 (2.5) | 8.8 (2.5)
HOMA-IR [Mean (Standard Deviation); unit: HOMA score] — There is no unit of measurement for HOMA-IR (Homeostatic model assessment - insulin resistance)
  HOMA score | 5.4 (3.0) | 4.6 (2.5) | 5.0 (2.8)
HOMA-beta cell [Mean (Standard Deviation); unit: percentage] | 64.9 (44.4) | 68.8 (63.1) | 66.9 (53.8)
Fasting Insulin [Mean (Standard Deviation); unit: microunits/milliters (uU/ml)] | 14.1 (7.8) | 12.6 (7.6) | 13.4 (7.7)
Fasting total-cholesterol [Mean (Standard Deviation); unit: micrograms/deciliter (mg/dL)] | 169.3 (27.7) | 169.9 (26.1) | 169.6 (26.9)
Fasting LDL-cholesterol [Mean (Standard Deviation); unit: micrograms/deciliter (mg/dL)] | 97.8 (22.3) | 96.2 (22.1) | 97.0 (22.2)
Fasting HDL-cholesterol [Mean (Standard Deviation); unit: micrograms/deciliter (mg/dL)] | 40.8 (6.3) | 44.2 (11.2) | 42.5 (8.8)
fasting triglycerides [Mean (Standard Deviation); unit: micrograms/deciliter (mg/dL)] | 153.1 (51.8) | 147.4 (59.8) | 150.3 (55.8)

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1C
Description: Change from baseline in hemoglobin A1C after 12 weeks of colesevelam or colesevelam plus sitagliptin treatments
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: percentage
Groups:
- Colesevelam Plus Sitagliptin: Colesevelam: Subjects were given 3.75 g colesevelam per day: 3 tablets (625mg each) with breakfast and 3 tablets (625mg each) with dinner for 12 weeks.
  Sitagliptin: Subjects were given 100mg sitagliptin per day: 1 tablet (100mg) with breakfast for 12 weeks.
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
percentage | 0.3 (1.2) | -0.1 (1.1)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

2. Secondary Outcome: Fasting Plasma C-peptide
Description: To evaluate the effect of treatments on plamsa C-peptide concentrations.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: picomoles (pmol)/Liter (L)
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 25
picomoles (pmol)/Liter (L) | 26 (217) | 103 (195)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

3. Primary Outcome: Fasting Plasma Glucose
Description: Change from baseline in fasting plasma glucose concentrations after 12 weeks of colesevelam or colesevelam plus sitagliptin treatments.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: millimoles (mmol)/Liter (L)
Groups:
- Colesevelam Plus Sitagliptin: Colesevelam: subjects were given 3.75 g colesevelam per day: 3 tablets (625mg each) with breakfast and 3 tablets (625mg each) with dinner for 12 weeks.
  Sitagliptin: Subjects were given 100 mg sitagliptin per day: 1 tablet (100mg) with breakfast for 12 weeks.
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
millimoles (mmol)/Liter (L) | -0.8 (2.1) | -0.6 (2.3)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effects between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

4. Secondary Outcome: Fasting Plamsa Glucagon
Description: To evaluate the effect of treatments on plasma glucagon concentrations.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: picograms (pg)/milliliter (ml)
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
picograms (pg)/milliliter (ml) | 1 (22) | 0 (17)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

5. Secondary Outcome: Fasting Active Plasma Glucagon Like-Peptide 1 (GLP-1)
Description: To evaluate the effect of treatments on plasma GLP-1 concentrations.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/L | 2.4 (4.2) | 2.8 (8.4)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

6. Secondary Outcome: Fasting Plasma Total Glucose-dependent Insulinotropic Peptide (GIP)
Description: To evaluate the effect of treatments on plasma Glucose-dependent Insulinotropic Peptide (GIP) concentrations.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/L | 1.8 (8.5) | -1.3 (3.4)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; unpaired t-test

7. Primary Outcome: Fasting Endogenous Glucose Production
Description: Change from baseline in fasting endogenous glucose production after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatment
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: micromoles (umol) per kg FFM per min
Groups:
- Colesevelam Plus Sitagliptin: Colesevelam: Subjects were given 3.75 g colesevelem per day: 3 tablets (625mg each) with breakfast and 3 tablets with dinner for 12 weeks.
  Sitagliptin: In addition subjects were given 100mg sitagliptin per day. Subjects were given 1 tablet (100mg) with breakfast for 12 weeks.
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
micromoles (umol) per kg FFM per min | 1.0 (4.4) | 1.0 (3.3)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Treament difference in fasting EGP between the 2 groups were compared; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

8. Primary Outcome: Fasting Gluconeogenesis
Description: Change from baseline in fasting gluconeogenesis after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatment
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: umol per kilogram (kg) FFM per min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
umol per kilogram (kg) FFM per min | 0.2 (1.5) | -0.3 (1.3)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between groups was evaluated; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

9. Primary Outcome: Fasting Glycogenolysis
Description: Change from baseline in fasting glycogenolysis after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatment
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: umol per kg Fat-Free Mass (FFM) per min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
umol per kg Fat-Free Mass (FFM) per min | 0.8 (3.6) | 1.7 (3.0)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between groups was evaluated; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired ttest

10. Primary Outcome: Fasting Plasma Glucose Clearance
Description: Change from baseline in fasting plasma glucose clearance after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatments.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: ml per kg FFM per minute (min)
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
ml per kg FFM per minute (min) | 0.30 (0.35) | 0.27 (0.41)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

11. Primary Outcome: Appearance Rate of Oral Glucose
Description: Change from baseline in appearance rate of oral glucose after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatments
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: umol per kg per min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
umol per kg per min | 118 (613) | -244 (464)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p = 0.01, t-test, 2 sided; unpaired t-test

12. Primary Outcome: Postprandial Endogenous Glucose Production
Description: Change from baseline in postprandial endogenous glucose production after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatments
  Mean value was calculated using all results measured between 10 and 300 min post meal.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: umol per kg per min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 25 | 26
umol per kg per min | -0.1 (2.0) | -0.2 (1.5)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; differerences in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

13. Primary Outcome: Postprandial Rate of Total Glucose Disposal Area Under the Curve (AUC)
Description: Change from baseline in postprandial rate of total glucose disposal (AUC) after 12 weeks of colesevelam alone or colesevelam plus sitagliptin treatments
  AUC was calculated by the trapezoid method using all results measured between 0 and 300 min during the meal tolerance test.
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: umol per kg per min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 25 | 26
umol per kg per min | -10 (914) | -256 (627)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

14. Primary Outcome: Whole-body Glycolytic Disposal of Oral Glucose
Description: Change in baseline in whole-body glycolytic disposal of oral glucose after 12 weeks of colesevelam alone or colesevelam plus glucose treatments
Time Frame: baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: Percent of Load
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 25 | 26
Percent of Load | 4 (6) | 2 (6)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

15. Primary Outcome: Postprandial Glucose (AUC)
Description: Comparison between baseline and 12 weeks values of postrandial glucose (AUC).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: millimoles (mmol)/l x min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 25 | 26
millimoles (mmol)/l x min | -1.1 (2.6) | -1.5 (2.8)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

16. Secondary Outcome: Fasting Insulin
Description: To evaluate the effect of treatments on fasting insulin concentrations
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/L
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/L | 6 (38) | 12 (36)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

17. Secondary Outcome: Postprandial Insulin (AUC)
Description: To evaluate the effect of treatments on postprandial insulin (AUC)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/l x min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/l x min | -13 (118) | 40 (73)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; unpaired t-test

18. Secondary Outcome: Postprandial C-peptide (AUC)
Description: To evaluate the effect of treatments on postprandial C-peptide (AUC)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/l x min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/l x min | 30 (390) | 193 (367)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; unpaired t-test

19. Secondary Outcome: Postprandial Active GLP-1 (AUC)
Description: To evaluate the effects of treatments on postprandial active GLP-1 (AUC)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/l x min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/l x min | 1.8 (7.9) | 6.6 (4.9)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; unpaired t-test

20. Secondary Outcome: Postprandial Total GIP (AUC)
Description: To evaluate the effects of treatment on postprandial total GIP (AUC)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: pmol/l x min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
pmol/l x min | -2 (6) | -5 (7)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p < 0.01, t-test, 2 sided; unpaired t-test

21. Secondary Outcome: Postprandial Glucagon (AUC)
Description: To evaluate the effects of treatment on postprandial glucagon (AUC)
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: picograms (pg)/milliter (ml) x min
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Number analyzed (Participants) | 24 | 26
picograms (pg)/milliter (ml) x min | -7 (15) | -4.7 (11)
Statistical Analysis 1: Comparison: Colesevelam vs Colesevelam Plus Sitagliptin; Difference in treatment effect between the 2 groups; Test type: Superiority or Other; p > 0.05, t-test, 2 sided; unpaired t-test

ADVERSE EVENTS:
Arm/Group | Colesevelam | Colesevelam Plus Sitagliptin
Serious Adverse Events (participants affected / at risk) | 0/31 | 0/30
Other Adverse Events (participants affected / at risk) | 1/31 | 1/30
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Colesevelam (N=31) | Colesevelam Plus Sitagliptin (N=30)
Tingling sensation in lower extremities (Nervous system disorders) | 1 (1) | 0 (0) — Subject complained of tingling sensation in lower extremities accompanied by headache and dry mouth.
Non-related Adverse Event (General disorders) | 0 (0) | 1 (1) — Subject withdrawn due to a non-related adverse event

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes